CLINICAL TRIAL: NCT06771739
Title: Preventing Financial Adversity Among Early-Stage Cancer Patients Through Unrestricted Cash (PAYMENT) Pilot Study
Brief Title: A Pilot Unrestricted Payment Program for Early-stage Cancer Patients: the PAYMENT Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1124982; NCI-2024-10341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UG1CA189974 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-06

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (high payment schedule) (Experimental): Patients receive a $1000 preloaded cash card once monthly for 3 months.
  Interventions: Other: Electronic Health Record Review; Other: Interview; Other: Support; Other: Survey Administration
- Arm B (low payment schedule) (Active Comparator): Patients receive a $100 preloaded cash card once monthly for 3 months.
  Interventions: Other: Electronic Health Record Review; Other: Interview; Other: Support; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
Other: Support — Receive $1000 preloaded cash card
  Other Names: Supportive - procedure intent
  Arms: Arm A (high payment schedule)
Other: Support — Receive $100 preloaded cash card
  Other Names: Supportive - procedure intent
  Arms: Arm B (low payment schedule)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether an unrestricted cash payment program can be used to improve financial and clinical outcomes in early-stage cancer patients with financial concerns. A cancer diagnosis can have poor financial outcomes, and the cost of cancer treatment can lead to high medical debt and financial hardships for the patient and family. Financial hardship during cancer treatment is associated with adverse outcomes including poorer quality of life, lower treatment compliance, more aggressive use of hospital-based care, and worse survival. Newly diagnosed cancer patients with financial concerns may avoid treatment entirely so that they can continue to work and maintain income, provide for their families, or pay rent. An unrestricted cash payment program provides patients with a preloaded cash card once monthly. The patients can choose what to use the card to pay for and may include items like food, rent, or utilities. This provides a period of guaranteed income for the patients and may prevent them from falling into poverty and improve financial and clinical outcomes.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive a $1000 preloaded cash card once monthly for 3 months.

ARM B: Patients receive a $100 preloaded cash card once monthly for 3 months.

After completion of study intervention, patients are followed up 3 months and 6 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Ability to understand English
* Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Within 90 days of a non-metastatic or early-stage solid tumor receiving or rescheduled to receive treatment in the neoadjuvant, adjuvant or definitive setting for curative intent. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Current cancer patient at PeaceHealth (Southwest Medical Center or St. Joes)
* Not current Medicaid enrollee
* Not enrolled in hospice
* Screens positive for financial fragility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant enrollment | Up to 1 year
  Feasibility will be measured by participant enrollment (percent enrolled versus [vs.] approached). The study will be considered feasible to implement if 60% or more of approached patients enroll.
Time to accrue 20 patients | Up to 1 year
  Feasibility will be measured by the time in months to accrue 20 patients. The study will be considered feasible if accrual is reached by 6 months.
Dropout rate | Up to 1 year
  Feasibility will be measured by dropout during study period. The study will be considered feasible to implement if less than 20% of patients drop out. Will be able to estimate a drop-out rate of 20% to within a 95% confidence interval of +/- 18%.
Survey completion rate | Up to 1 year
  Feasibility will be measure by rates of survey completion. The study will be considered feasible to implement if survey completion is 90% or greater.

SECONDARY OUTCOMES:
Financial hardship | Baseline, 3 and 6- months post randomization
  Will assess whether patient self-reports one or more of the following: new debt (relative to baseline), income decline of 20% or more, loans from family/friends to pay for cancer treatment, selling/refinancing primary home, >= 2 months missed rent or mortgage payments, evictions. May adjust either the methods for assessing financial hardship (e.g. using credit reports rather than surveys) or the endpoint itself based on observed survey completion rate and incidence of each endpoint.
Treatment nonadherence | Baseline, 3 and 6- months post randomization
  Will assess whether patient self reports they did or did not skip medication doses or refuse/decline recommended therapy due to cost concerns. Evidence of treatment completion vs. missed treatments/appointments using data from electronic medical record captured by research assistant.
Unplanned emergency department (ED)/hospital admissions | Baseline, 3 and 6- months post randomization
  All instances of ED visits and hospital stays (including reason for visit) will be abstracted from patients' medical records. The study team will categorize visits as anticipated (for chemotherapy or planned procedure) vs. unanticipated (complication or treatment side effect).
Food and housing insecurity | Baseline, 3 and 6- months post randomization
  Will be assessed using items 1 through 4 of the 10-item Health-Related Social Needs Screening Tool from Centers for Medicare and Medicaid Services.
Quality of life | Baseline, 3 and 6- months post randomization
  Will be assessed using the composite score from the European Quality of Life Five Dimension Index (scored 0-100). A 6-point score change is considered clinically meaningful in United States cancer populations.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Shankaran, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No